CLINICAL TRIAL: NCT06963203
Title: Thyroidectomy for Graves' Disease or Amiodarone-induced Thyrotoxicosis: Is it Still Necessary to Achieve a Preoperative Euthyroid State? - A Prospective Observational Multicenter European Study (GRATES)
Brief Title: Thyroidectomy for Graves' Disease or Amiodarone-induced Thyrotoxicosis
Acronym: GRATES
Status: Recruiting | Type: Observational
Sponsor: Andrea Goldmann (Other)
Collaborators: Spital Männedorf (Unknown); Spital Limmattal Schlieren (Other); Centre Hospitalier Universitaire Vaudois (Other); Ospedale Regionale di Mendrisio (Other); Cantonal Hospital of St. Gallen (Other); Cantonal Hosptal, Baselland (Other); St. Claraspital AG (Other); University Hospital, Geneva (Other); Insel Gruppe AG, University Hospital Bern (Other); ASZ Aalst (Other); University Hospital Virgen de las Nieves (Other); University of Nancy (Other); Hospital Costa del Sol (Other); Evgenidion Hospital Athens, Greece (Unknown)
Responsible Party: Sponsor-Investigator, Andrea Goldmann, Fellow of the European Board of Surgery (FEBS) - Endocrine Surgery, Schwerpunkt Viszeralchirurgie, FMH Chirurgie, Kantonsspital Winterthur Klinik für Viszeral- und Thoraxchirurgie Stv. Chefärztin und Stv. Klinikleiterin, Teamleiterin Endokrine Chirurgie, Kantonsspital Winterthur KSW
Organization: Kantonsspital Winterthur KSW (Other)
Other Study IDs: BASEC Nr 2024-01766
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Graves Disease; Amiodarone-Induced Thyrotoxicosis; Thyroidectomy
Keywords: GRATES; GRATE Study; thyreotoxicosis; euthyreoidism; Thyroid storm
MeSH Terms: conditions — Graves Disease; Thyroid Crisis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- euthyreoid: Patients undergoing thyroidectomy in a euthyreoid state.
- non-euthyreoid: Patients undegoing thyroidectomy in a non-euthyreoid state.

SUMMARY:
The goal of this observational study is to learn about the potential differences in morbidity of thyroidectomy (removal of the thyroid gland) depending on the preoperative hormonal status. The main question it aims to answer is:

Do patients undergoing thyroidectomy for thyreotoxicosis (thyroid hyperfunction) due to Graves' disease or Amiodarone induced thyreotoxicosis have comparable complication rates depending on their thyroid metabolic status prior or during the procedure.

The data from participants undergoing a thyroidectomy at one of the study sites will be prospectively registered in the EUROCRINE registry, including an add-on module for additional study specific routine data. The operation itself, the preoperative or postoperative treatments are not altered in any way.

DETAILED DESCRIPTION:
Background:

Thyrotoxicosis is the clinical condition associated with excessive thyroid hormone activity, usually due to inappropriately high levels of circulating thyroid hormones. The clinical presentation is variable, ranging from asymptomatic to life-threatening 'thyroid storm'. Symptoms include weight loss, heat intolerance and palpitations. Thyrotoxicosis can result from diffuse alterations of the thyroid gland, such as Graves' disease and Amiodarone-induced thyrotoxicosis (AIT). This poses a considerable challenge across multiple medical specialties, spanning endocrinology, cardiology, and anesthesiology.

Graves' disease is a widespread endocrine disorder that affects approximately 1% of the population. Treatment strategies vary based on clinical presentation and patient preferences, with options ranging from medical management to thyroidectomy. Amiodarone is a class III antiarrhythmic drug used to treat supraventricular and ventricular arrhythmias, and to maintain sinus rhythms after cardioversion of atrial fibrillation. Its prescription has become more common in recent decades. However, the medication comes with the risk of precipitating severe thyrotoxicosis, which, if left untreated, can be fatal. Discontinuing the medication may not always be feasible.

Under medical treatment for thyrotoxicosis (using thionamides or glucocorticoids), attaining euthyroidism can frequently be challenging to achieve, prompting consideration of definitive treatment through thyroidectomy.

Thyroidectomy for Graves' disease or AIT presents unique disease-specific challenges, potentially resulting in elevated perioperative complication rates when compared to other indications. According to current guidelines, it is recommended to attain a euthyroid state prior to surgery to mitigate perioperative risks, despite the inconclusive evidence supporting this approach. Nevertheless, data from retrospective studies show that between 21-51% of patients undergo surgery when euthyroidism is not stable or cannot be achieved.

The EUROCRINE® registry offers a valuable opportunity to assess the morbidity linked to thyroidectomy for Graves' disease and AIT, considering both euthyroid and hyperthyroid states. This prospective, observational study aims to refine surgical protocols and inform updates to existing guidelines, thereby advancing the management of thyroidectomy for Graves' disease and AIT.

Objectives:

The aim of this study is to explore potential differences in the morbidity of thyroidectomy for Graves' disease and AIT based on thyroid metabolic status prior to or during the procedure. The study hypothesis is that there will be no significant differences in relevant complication rates, such as transient and permanent nerve palsy, transient and permanent hypoparathyroidism, reoperation, severe adverse intraoperative cardiac events, or the onset of a "thyroid storm".

If this hypothesis is confirmed, patients with Graves' disease and AIT who are scheduled for thyroidectomy would no longer need to wait to reach a state of euthyroidism. This would streamline preoperative assessments and expedite surgical planning, leading to reduced costs and shorter waiting times, and minimizing exposure to dangerous and excessive levels of thyroxine.

The primary endpoint is the relevant complication rate in both groups: transient and permanent nerve palsy, transient and permanent hypoparathyroidism, reoperation for postoperative haemorrhage, and occurrence of a "thyroid storm".

The secondary endpoints are results of other complications, duration of surgery, estimated blood loss, intraoperative tachycardia, length of hospital stay, ICU monitoring, preoperative medications, use of autofluorescence, angiofluorescence, and neuromonitoring, preoperative calcium and/or vitamin D supplementation, clinic volume.

Design:

The investigatiors are planning a prospective, observational, multicenter, multinational study based on the EUROCRINE® registry. Eurocrine® is an international endocrine surgical quality registry based in the EU. The project will be a Swiss national and multinational multicenter study.

Several other in Eurocrine® participating, international clinics have agreed to participate in the study. It is planned that a total of around 25 clinics in various European countries will take part in the study. In a first step, the participating centers in Switzerland will be opened.

The data will be entered prospectively into the online registry in encrypted form, which is the standard for the Eurocrine® registry. For the Eurocrine® registry itself a declaration of no objection has been issued in May 2017 for Switzerland (2017-00683). The clinics participating in the study do this part of the data entry unchanged from before. The participant can then be enrolled in the study via a my-Eurocrine add-on module and additional study-specific routine data can be collected directly in the Registry online platform. All variables, along with the study- specific variables, are systematically collected in the centers as a component of patient care, since these parameters are essential for treatment. The operation itself, the preoperative or postoperative treatments are not altered in any way. Information about postoperative complications will be registered at the Eurocrine® database as previously implemented.

Patients with Graves' disease or AIT can be included in this study and will be assigned to two groups. The investigators rely on free triiodothyronine (fT3) and free thyroxine (fT4) levels to assess functional status since the TSH level may not accurately reflect the patient's true functional status. Patients will be classified as uncontrolled if their levels of fT3 or fT4 are elevated, or as controlled (normal fT3 and fT4) immediately prior to surgery (normal ranges for all ages: fT4 12.0 - 22.0 pmol/l; fT3 3.1 - 6.8 pmol/l). The fT3 and fT4 tests will be conducted no more than one week before surgery. Consecutive patient enrolment is necessary to accurately reflect real clinical conditions. The standard variables are recorded as usual, with the addition of the study-specific variables (see CRF). All complications will be documented to evaluate the risk of surgery in both controlled and uncontrolled metabolic states.

For diagnosing patients with "thyroid storm", the investigators opted to utilize the established Japanese Association classification, which is deemed more suitable for clinical settings compared to the "Burch and Wartofsky" scale.

Origin of the data:

The investigators want to analyze data routinely collected in the clinical practice for adult, non- pregnant patients who underwent surgical management of Graves ' disease and AIT in different functional states. The variables are summarized in the CRF.

All data will be collected in the Eurocrine database with the standard module and an add-on specific variable my-Eurocrine module for study specific routine data. All participating sites will use the Eurocrine database and collect their data prospectively online and in a coded form. In the Eurocrine data registry, data is routinely recorded up to six months postoperatively in the event of complications occurring during treatment. This period also corresponds to that of the study project.

It is planned to run the study for 2 years and the study will start as soon as a positive ethical decision has been made. If enough patients have been enrolled before the end of the 2 years, the study will be stopped early.

Information and consent of participants:

The investigators will collect and analyze data routinely collected in clinical practice. The consent procedure at all Swiss sites are as followed:

Patients are informed through the documents entitled <General consent for the re-use of health-related data and samples for research purposes.>. All study patients provide approved informed consent for the further use of their medical records and tissue samples using the general document from the Hospital.

For clinics that do not have general consent, the Eurocrine consent form is used as standard (German and English versions available).

If a patient does not agree to the General Consent of the Swiss sites using the General Consent, but agrees to the use of data related to the thyroid disease and treatment, the patient can be enrolled in the study by signing the Eurocrine Consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) undergoing surgical treatment for Graves' disease or Amiodarone-induced thyrotoxicosis (AIT) with biochemically confirmed hyperthyroidism or on specific medication for the treatment of Graves' disease or AIT.
* Patients providing signed informed consent.

Exclusion Criteria:

* Children and minors (<18 years).
* Pregnant women.
* Patients unable or unwilling to provide informed consent due to language barriers or intellectual limitations.
* Patients undergoing concurrent parathyroidectomy for primary or secondary hyperparathyroidism, lymph node clearance, or redo surgery.
* Surgical procedures performed for other reasons than Graves' disease or AIT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, non- pregnant patients who underwent surgical management of Graves ' disease and AIT (Amiodarone induced thyreotoxicosis) in different functional states.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Complications | Day 0= intraoperative until last follow-up postoperatively (e.g. for the recovery from a nerve palsy)= through study completion, an average of 2 years
  transient and permanent nerve palsy, transient and permanent hypoparathyroidism, reoperation for postoperative hemorrhage, occurrence of a "thyroid storm"

SECONDARY OUTCOMES:
Other complications | From day 0= intraoperatively until last follow-up postoperatively (= through study completion, an average of 2 years)
  Any other intra- or postoperative complication.
Duration of Surgery | through study completion, an average of 2 years
  Time from start of the procedure until the end of the procedure
Estimated Blood Loss | During procedure
  Estimated amount of blood lost during the procedure.
Intraoperative Tachycardia | During the procedure
  Elevated heart rate during the procedure
Lenght of Hospital Stay | From day 0= intraoperatively until last follow-up postoperatively (= through study completion, an average of 2 years)
  Duration a patient remained at the hospital when undergoing the procedure. Date from surgery until discharge.
ICU monitoring | From day 0= intraoperatively until last follow-up postoperatively (= through study completion, an average of 2 years)
  Was the patient monitored at the ICU (for any reason) during the postoperative period.
Preoperative Medications | From day 0= intraoperatively and prior records (after study inclusion=baseline)
  What medications did patients have prior to/when undergoing the procedure
Autofluorescence | During the procedure
  Intraoperative use of autofluorescence for the identification of the parathyroid glands.
Angiofluorescence | During the procedure
  Intraoperative use of angiofluorescence for the identification of the parathyroid glands.
Neuromonitoring | During the procedure
  Ude of a neuromonitoring device during the procedure
Preoperative Calcium or Vitamin D supplementation | Preoperative Study Period
  Indication wheter a patient received preoperative Vitamin D or Calcium as supplementation
Clinic Volume | Baseline
  Number of thyroid surgeries annually performed at a clinic in order to categorize participating hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Goldmann, MD, Principal Investigator — Kantonsspital Winterthur KSW
Locations (15):
- OLV Ziekenhuis, Aalst, Belgium
- Universite de Lorraine, Cru Nancy, Nancy, France
- Evgenidion Hospital Athens, Athens, Greece
- Spain (2):
  - Universitario Virgen de las Nieves, Granada
  - Hospital Costa del Sol, Marbella
- Switzerland (10):
  - Kantonsspital Winterthur, Zurich, Winterthur
  - Clarunis St. Clara Spital, Basel
  - Universitätsspital Bern, Inselspital, Bern
  - University Hospitals of Geneva, Geneva
  - University Hospital of Lausanne CHUV, Lausanne
  - Kantonsspital Basel Land, Liestal
  - Spital Männedorf, Männedorf
  - Ospedale Regionale di Mendrisio, Mendrisio
  - HOCH Kantonsspital St. Gallen, Sankt Gallen
  - Spital Limmattal, Schlieren

IPD SHARING:
Plan to Share IPD: Undecided
International multicenter study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT06963203/Prot_SAP_000.pdf